CLINICAL TRIAL: NCT04818437
Title: Effect of Core Stability Exercises and Balance Training in Postural Control Among Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/19/1012 Hunza Zulfiqar
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Core stability; Postural Control; Pediatric Berg balance scale
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance training (Experimental): Balance training
  1. Trunk, head, and upper limbs rotation from kneeling.
  2. Upper limbs flexion and extension with simultaneous head movement from kneeling.
  3. Pelvic bridging followed by raising one lower limb and extending knee.
  4. Lifting opposite upper and lower limbs from Quadruped position.
  6-Heel and toe raises, alternate rising ofthe right and left feet above the floor, and tandem standing. 7-Weight shifting forward. backward, sideward, and diagonally with eyes opened and eyes closed
  Interventions: Other: BALANCE TRAINING
- Core stability exercise (Active Comparator): Core stability exercises:
  1. Abdominal bracing while lying in supine position.
  2. Abdominal bracing with heel slide while lying in supine position.
  3. Abdominal bracing with Leg lifts while lying in supine position.
  4. Abdominal bracing with bridging while lying in supine position.
  5. Abdominal bracing while Standing 6-Abdominal bracing while walking.
  7-Quadra pod arm lifts with bracings while Quadra pod position. 8-Quadra pod alternate arm and leg lifts with bracing while Quadra pod position. 9-Side plank with knee flexion while side lying. 10-Side plank with knee extension while side lying.
  Interventions: Other: CORE STABILITY EXERCISES

INTERVENTIONS:
Other: BALANCE TRAINING — Trunk, head, and upper limbs rotation from kneeling. 2- Upper limbs flexion and extension with simultaneous head movement from kneeling. 3-Pelvic bridging followed by raising one lower limb and extending knee. 4-Lifting opposite upper and lower limbs from Quadruped position. 6-Heel and toe raises, alternate rising of he right and left feet above the floor, and tandem standing. 7-Weight shifting forward. backward, sideward, and diagonally with eyes opened and eyes closed
  Arms: Balance training
Other: CORE STABILITY EXERCISES — 1. Abdominal bracing while lying in supine position.
  2. Abdominal bracing with heel slide while lying in supine position.
  3. Abdominal bracing with Leg lifts while lying in supine position.
  4. Abdominal bracing with bridging while lying in supine position.
  5. Abdominal bracing while Standing.-Abdominal bracing while walking.
  7-Quadra pod arm lifts with bracings while Quadra pod position. 8-Quadra pod alternate arm and leg lifts with bracing while Quadra pod position. 9-Side plank with knee flexion while side lying. 10-Side plank with knee extension while side lying
  Arms: Core stability exercise

SUMMARY:
Children with Down syndrome often present with problems of posture & balance and mobility. Balance training is an important component of physical activity interventions, with growing evidence that it can be beneficial for children with DS.

Objective: To determine the effect core stability exercises and balance training in postural control among Down syndrome.

DETAILED DESCRIPTION:
This study was a randomized clinical trail. Children with Down Syndrome were determined on inclusion & exclusion criteria. Children with Down syndrome were arbitrarily allocated into two groups with ages ranged from 5 to 17 years. The sample size was 20 patients. They were assigned randomly into two groups. Group 1 received balance training and Group 2 received core stability exercises. The duration of treatment was 6 weeks. Data is collected from Comprehensive Rehabilitation center Chakwal Postural stability was evaluated pre and post treatment by pediatric berg balance scale. Values which were obtained after this intervention were analyzed for any change using SPSS

ELIGIBILITY:
Inclusion Criteria:

* Trisomy 21 by genetic karyotype
* A confirmed diagnosis of Down syndrome by a paediatric neurologist, having no neurological or mobility disorders,
* independent standing and walking abilities,
* Joint Laxity , low muscle tone and psychomotor development deficits
* Normal vision and hearing

Exclusion Criteria:

* A history of congenital heart defects and orthopedic
* surgery in the past year and severe mental retardation.
* Seizure
* Severe visual or auditory disturbances,
* Weight less than the 3rd percentile of Down syndrome
* Multiple sclerosis or epilepsy

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg balance scale | 2 months
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in CP children . The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Binash afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsakhawi RS, Elshafey MA. Effect of Core Stability Exercises and Treadmill Training on Balance in Children with Down Syndrome: Randomized Controlled Trial. Adv Ther. 2019 Sep;36(9):2364-2373. doi: 10.1007/s12325-019-01024-2. Epub 2019 Jul 12. PMID 31301057
- [Background] Eid MA, Aly SM, Huneif MA, Ismail DK. Effect of isokinetic training on muscle strength and postural balance in children with Down's syndrome. Int J Rehabil Res. 2017 Jun;40(2):127-133. doi: 10.1097/MRR.0000000000000218. PMID 28146007
- [Background] Zago M, Duarte NAC, Grecco LAC, Condoluci C, Oliveira CS, Galli M. Gait and postural control patterns and rehabilitation in Down syndrome: a systematic review. J Phys Ther Sci. 2020 Apr;32(4):303-314. doi: 10.1589/jpts.32.303. Epub 2020 Apr 2. PMID 32273655
- [Background] Sugimoto D, Bowen SL, Meehan WP 3rd, Stracciolini A. Effects of Neuromuscular Training on Children and Young Adults with Down Syndrome: Systematic Review and Meta-Analysis. Res Dev Disabil. 2016 Aug;55:197-206. doi: 10.1016/j.ridd.2016.04.003. Epub 2016 Apr 25. PMID 27123540
- [Background] Motealleh A, Mohamadi M, Moghadam MB, Nejati N, Arjang N, Ebrahimi N. Effects of Core Neuromuscular Training on Pain, Balance, and Functional Performance in Women With Patellofemoral Pain Syndrome: A Clinical Trial. J Chiropr Med. 2019 Mar;18(1):9-18. doi: 10.1016/j.jcm.2018.07.006. Epub 2019 Feb 10. PMID 31193229
- [Background] Maiano C, Hue O, Lepage G, Morin AJS, Tracey D, Moullec G. Do Exercise Interventions Improve Balance for Children and Adolescents With Down Syndrome? A Systematic Review. Phys Ther. 2019 May 1;99(5):507-518. doi: 10.1093/ptj/pzz012. PMID 31089706
- [Background] Capio CM, Mak TCT, Tse MA, Masters RSW. Fundamental movement skills and balance of children with Down syndrome. J Intellect Disabil Res. 2018 Mar;62(3):225-236. doi: 10.1111/jir.12458. Epub 2017 Dec 5. PMID 29205624
- [Background] Silva V, Campos C, Sa A, Cavadas M, Pinto J, Simoes P, Machado S, Murillo-Rodriguez E, Barbosa-Rocha N. Wii-based exercise program to improve physical fitness, motor proficiency and functional mobility in adults with Down syndrome. J Intellect Disabil Res. 2017 Aug;61(8):755-765. doi: 10.1111/jir.12384. Epub 2017 Jun 6. PMID 28585394
- [Background] Pena GM, Pavao SL, Oliveira MFP, Godoi D, de Campos AC, Rocha NACF. Dual-task effects on postural sway during sit-to-stand movement in children with Down syndrome. J Intellect Disabil Res. 2019 Jun;63(6):576-586. doi: 10.1111/jir.12599. Epub 2019 Jan 28. PMID 30687997
- [Background] Saquetto MB, Pereira FF, Queiroz RS, da Silva CM, Conceicao CS, Gomes Neto M. Effects of whole-body vibration on muscle strength, bone mineral content and density, and balance and body composition of children and adolescents with Down syndrome: a systematic review. Osteoporos Int. 2018 Mar;29(3):527-533. doi: 10.1007/s00198-017-4360-1. Epub 2018 Jan 12. PMID 29330572